CLINICAL TRIAL: NCT02609256
Title: Stereotactic Infarct Tissue Aspiration (SITA) for Malignant Infarction of Middle Cerebral Artery
Brief Title: Stereotactic Infarct Tissue Aspiration for Malignant Infarction of Middle Cerebral Artery
Acronym: SMART
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director of Neurology Dept., General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k(2015)32
Record Dates: First submitted 2015-11-11; First posted 2015-11-20 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Middle Cerebral Artery Infarction
Keywords: Intracranial hypertension; cerebral herniation; Stereotactic infarct tissue aspiration; fatality; disability
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Intracranial Hypertension | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stereotactic infarct tissue aspiration (Experimental): Patients receive the stereotactic infarct tissue aspiration 24-48 hours after cerebral infarction beside medical therapy.
  Interventions: Procedure: Stereotactic infarct tissue aspiration; Other: Medical therapy
- Medical therapy (Sham Comparator): osmotic therapy with mannitol and glycerol fructose，anti-platelet treatment, statins, and other symptomatic treatments such as controlling blood pressure, blood sugar, and infection, and tracheal intubation or incision, etc;
  Interventions: Other: Medical therapy

INTERVENTIONS:
Procedure: Stereotactic infarct tissue aspiration — The patient posed supine position to expose local skin and puncture point was located at 6.5 cm behind the hairline of the lesion side, and 5.0 cm lateral of midline. After routine skin preparation and disinfection, 5% lidocaine 2-5 ml was injected for local anesthesia. The skin was cut to expose periosteum by a scalpel. After skull was vertically drilled through with a 6mm diameter hole, a sterile tube with a needle in tube was put about 8 cm into centrum semiovale. The needle was put out and about 50ml necrosis brain tissue was aspirated by a 20 ml syringe. The tube was fixed into the skin about 2 cm after subcutaneous tunnel, and connected to the drainage bag. Surgical area was sterilized and wrapped by sterile gauze bandage.
  Arms: Stereotactic infarct tissue aspiration
Other: Medical therapy — osmotic therapy with mannitol and glycerol fructose，anti-platelet treatment, statins, and other symptomatic treatments such as controlling blood pressure, blood sugar, and infection, and tracheal intubation or incision, etc

SUMMARY:
Malignant middle cerebral artery infarction(MMCI) has a high rate of disability and mortality. At present, there is no effective treatment except for craniotomy decompression, but the controversy of the craniotomy decompression still exists. The project is a prospective, randomized, single center, open label, clinical controlled trail. The eligible patients for enrollment are as follows: (1) malignant cerebral artery infarction within 48h onset; (2) craniotomy decompression can not be performed due to the contraindications, or refused by the patient or relatives. The patients are randomly assigned into 2 groups: (1)Medical therapy group: receiving osmotic therapy with mannitol and glycerol fructose，anti-platelet treatment, statins, and other symptomatic treatments such as controlling blood pressure, blood sugar, and infection, tracheal intubation or incision, etc; (2) Stereotactic infarct tissue aspiration (SITA) group: on the basis of medical treatment, receiving minimally invasive aspiration of infarct tissue 24-48 hours after stroke attacked. This study is aimed at comparing the efficacy and safety of of SITA in patients with MMCI.

DETAILED DESCRIPTION:
Malignant middle cerebral artery infarction (MMCI) has a fatality rate of up to 80%, due to massive brain edema, increased intracranial pressure, and cerebral herniation. The herniation-induced death usually occured during the first week, despite aggressive osmotherapy with mannitol or hypertonic saline, sedation, and eventually hyperventilation, buffers, or hypothermia. A growing evidence show that decompression craniectomy (DC) can produce a significant reduction in mortality rate and an improvement in neurological outcome, but the controversy of the DC still exists. There is an urgent need to find a more effective treatment method. Given that brain tissue necrosis-induced edema and cerebral herniation is the key reason of fatality and disability of MMCI patients, the investigators argue that the reduction of cerebral tissue volume by stereotactic infarct tissue aspiration (SITA) is likely to reach the decompression effect similar to the DC. Recently, the investigators performed SITA in 2 MMCI patients who were qualified for decompressive craniectomy, but refused by patient relatives, and their neurological function significantly improved.

The project is a prospective, randomized, single center, open label, clinical controlled trail. The eligible patients for enrollment are as follows: (1)ages from 40 to 90 years old; (2) malignant cerebral artery infarction within 48h onset; (3) craniotomy decompression can not be performed due to the contraindications, or refused by the patient or relatives. The patients are randomly assigned into 2 groups: (1) Medical therapy group: receiving osmotic therapy with mannitol and glycerol fructose，anti-platelet treatment, statins, and other symptomatic treatments such as controlling blood pressure, blood sugar, and infection, and tracheal intubation or incision, etc; (2) SITA group: receiving minimally invasive aspiration of infarct tissue 24-48 hours after stroke attacked on the basis of medical treatment. This study is aimed at comparing the efficacy and safety of of SITA in patients with MMCI.

ELIGIBILITY:
Inclusion Criteria:

1. ages from 40 to 90
2. within 48 hours of onset
3. brain imaging confirmed malignant middle cerebral artery infarction (DWI+MRA)
4. infarction volume > 145ml
5. craniotomy decompression can not be performed due to the contraindications, or refused by the patient or relatives
6. signed informed consent.

Exclusion Criteria:

1. hemorrhagic stroke
2. severe infection or severe disfunction of liver, kidney, hematopoietic system, endocrine system and other serious diseases
3. other clinical trials within 3 months
4. a negative attitude towards SITA by patient or relatives
5. other conditions not eligible for the trail judged by the researchers.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale(mRS) 0-3 vs mRS 4-6 | 90±7days

SECONDARY OUTCOMES:
National Institute of Health stroke scale(NIHSS) | 14±2days
  NIHSS score improvement
Mean survival time | 1 year
death due to any reasons | 90±7days
mRS 0-4 compared with mRS 5 or 6 | 90±7days

OTHER OUTCOMES:
The number of Local hemorrhage cases | 14±2 days
The number of intracranial hemorrhage cases | 14±2 days
Major cardiovascular events | during the surgery
The number of intracranial infection cases | 14±2 days
The number of Local infection cases | 14±2 days

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen Jing Qiu, PhD, Study Chair — Director
Locations (1):
- General hospital of shenyang military region, Shenyang, Liaoning, China

REFERENCES:
- [Background] van Middelaar T, Richard E, van der Worp HB, van den Munckhof P, Nieuwkerk PT, Visser MC, Stam J, Nederkoorn PJ. Quality of life after surgical decompression for a space-occupying middle cerebral artery infarct: A cohort study. BMC Neurol. 2015 Aug 28;15:156. doi: 10.1186/s12883-015-0407-0. PMID 26311142
- [Background] Hofmeijer J, Amelink GJ, Algra A, van Gijn J, Macleod MR, Kappelle LJ, van der Worp HB; HAMLET investigators. Hemicraniectomy after middle cerebral artery infarction with life-threatening Edema trial (HAMLET). Protocol for a randomised controlled trial of decompressive surgery in space-occupying hemispheric infarction. Trials. 2006 Sep 11;7:29. doi: 10.1186/1745-6215-7-29. PMID 16965617
- [Background] Neugebauer H, Heuschmann PU, Juttler E. DEcompressive Surgery for the Treatment of malignant INfarction of the middle cerebral arterY - Registry (DESTINY-R): design and protocols. BMC Neurol. 2012 Oct 2;12:115. doi: 10.1186/1471-2377-12-115. PMID 23031451
- [Background] Raffiq MA, Haspani MS, Kandasamy R, Abdullah JM. Decompressive craniectomy for malignant middle cerebral artery infarction: Impact on mortality and functional outcome. Surg Neurol Int. 2014 Jun 26;5:102. doi: 10.4103/2152-7806.135342. eCollection 2014. PMID 25101197
- [Background] Hatefi D, Hirshman B, Leys D, Lejeune JP, Marshall L, Carter BS, Kasper E, Chen CC. Hemicraniectomy in the management of malignant middle cerebral artery infarction: Lessons from randomized, controlled trials. Surg Neurol Int. 2014 May 15;5:72. doi: 10.4103/2152-7806.132589. eCollection 2014. No abstract available. PMID 24991475
- [Background] Vahedi K, Vicaut E, Mateo J, Kurtz A, Orabi M, Guichard JP, Boutron C, Couvreur G, Rouanet F, Touze E, Guillon B, Carpentier A, Yelnik A, George B, Payen D, Bousser MG; DECIMAL Investigators. Sequential-design, multicenter, randomized, controlled trial of early decompressive craniectomy in malignant middle cerebral artery infarction (DECIMAL Trial). Stroke. 2007 Sep;38(9):2506-17. doi: 10.1161/STROKEAHA.107.485235. Epub 2007 Aug 9. PMID 17690311
- [Background] Simard JM, Sahuquillo J, Sheth KN, Kahle KT, Walcott BP. Managing malignant cerebral infarction. Curr Treat Options Neurol. 2011 Apr;13(2):217-29. doi: 10.1007/s11940-010-0110-9. PMID 21190097
- [Background] Juttler E, Unterberg A, Woitzik J, Bosel J, Amiri H, Sakowitz OW, Gondan M, Schiller P, Limprecht R, Luntz S, Schneider H, Pinzer T, Hobohm C, Meixensberger J, Hacke W; DESTINY II Investigators. Hemicraniectomy in older patients with extensive middle-cerebral-artery stroke. N Engl J Med. 2014 Mar 20;370(12):1091-100. doi: 10.1056/NEJMoa1311367. PMID 24645942